CLINICAL TRIAL: NCT00682305
Title: Allogeneic Stem Cell Transplantation With Treosulfan, VP-16 and Cyclophosphamide for Patients With Acute Lymphoblastic Leukemia (ALL) Not Eligible for TBI-containing Conditioning Regimen: A Phase II-study
Brief Title: Allogeneic Stem Cell Transplantation (SCT) With Treosulfan, VP-16 and Cyclophosphamid for Patients With Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TreoALL
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Hematopoeitic Stem Cell Transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-Arm (Other): Single-Arm
  Interventions: Procedure: Hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Hematopoietic stem cell transplantation — conditioning regimen:
  * day -7: 12g/m^2 Treosulfan
  * day -6: 12g/m^2 Treosulfan
  * day -5: 12g/m^2 Treosulfan
  * day -4: 30mg/kg BW Etoposide
  * day -3: 20mg/kg ATG Fresenius (OPTIONAL), 60mg/kg BW Cyclophosphamide
  * day -2: 20mg/kg ATG Fresenius (OPTIONAL), 60mg/kg BW Cyclophosphamide
  * day -1: 20mg/kg ATG Fresenius (OPTIONAL)
  * day 0: SCT

SUMMARY:
The present study is a multicenter, prospective phase II-study investigating the combination of treosulfan, etoposide, and cyclophosphamide as conditioning regimen for patients with acute lymphoblastic leukemia who are not eligible for a TBI-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia in first or subsequent complete remission
* Indication for allogeneic stem cell transplantation according to the actual protocol of the German Acute Lymphoblastic Leukemia Study Group
* Patient's age: 18-65 years
* HLA-identical or compatible related or unrelated donor (HLA-A, HLA-B, HLA-C, HLA-DRB1 and HLA-DQB1) (one antigen-mismatch allowed)
* Not eligible for total-body irradiation due to one of the following reasons:

  * prior radiation of the spine > 30 Gy
  * prior radiation of the mediastinum > 30 Gy
  * severe pulmonary infection during induction chemotherapy
  * DLCO > 50%
* Patient's wishing to avoid total-body irradiation as conditioning regimen
* Patient's written informed consent
* Women and men capable of reproduction must agree to use highly effective methods of contraception until six months after treatment termination. For men: vasectomy, sexual abstinence, or partner is using hormonal IUD, implants, injectables, oral hormonal contraceptives or is surgically sterilized. For women: hormonal IUD, implants, injectables, sexual abstinence, surgical sterilization, vasectomised partner

Exclusion Criteria:

* No complete remission at time of registration
* Severe irreversible renal, hepatic, pulmonary or cardiac disease, such as

  * total bilirubin, SGPT or SGOT > 3 times upper the normal level
  * Left ventricular ejection fraction < 30%
  * Creatinine clearance < 30 ml/min
  * DLCO < 35% and/ or receiving supplementary continuous oxygen
* Positive serology HIV
* Pregnant or lactating women
* Severe florid infection
* Experienced hypersensitivity against cyclophosphamid, etoposide, or treosulfan
* Cystitis
* Obstructive renal function
* Participation in any other clinical drug trial
* Serious psychiatric or psychological disorders
* Progressive invasive fungal infection at time of registration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2013-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of engraftment at day +28 and non-relapse mortality at day +100 and at 1 year after SCT | 1 year after SCT

SECONDARY OUTCOMES:
*Incidence of aGvHD on day +100/ cGvHD at 1 and 2 yrs after SCT/ relapse at 2 yrs after SCT *Toxicity *Disease-free survival at 2 yrs after SCT *overall survival at 2 yrs. after SCT | 2 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kroeger, Prof. Dr., Principal Investigator — University Medical Center Hamburg-Eppendorf, Department for Stem Cell Transplantation
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Kroger N, Bornhauser M, Stelljes M, Pichlmeier U, Trenschel R, Schmid C, Arnold R, Martin H, Heinzelmann M, Wolschke C, Meyer RG, Bethge W, Kobbe G, Ayuk F, Gokbuget N, Holzer D, Zander A, Beelen D. Allogeneic stem cell transplantation after conditioning with treosulfan, etoposide and cyclophosphamide for patients with ALL: a phase II-study on behalf of the German Cooperative Transplant Study Group and ALL Study Group (GMALL). Bone Marrow Transplant. 2015 Dec;50(12):1503-7. doi: 10.1038/bmt.2015.202. Epub 2015 Sep 14. PMID 26367236